CLINICAL TRIAL: NCT04981132
Title: Investigation of the Effectiveness of Pain and Exercise Training With Telerehabilitation Method in Patients With Low Back Pain Caused by Lumbar Facet Joint Arthrosis
Brief Title: Effectiveness of Pain and Exercise Training With Telerehabilitation on Lumbar Facet Joint Arthrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Begüm Okudan, MSc. Pt, Okan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0366
Record Dates: First submitted 2021-06-21; First posted 2021-07-28 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Facet Joint Arthrosis; Low Back Pain
Keywords: facet joint arthrosis; low back pain; exercise; education; telerehabilitation
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Education+Exercise Group (Experimental): Group 1: Patients will have 15 minutes of pain neuroscience education (PNE) and 30 minutes of progressive therapeutic exercise training (PTE) with the telerehabilitation method.
  Interventions: Behavioral: Pain Neuroscience education + Progressive therapeutic exercise training
- Exercise group (Experimental): Group 2: Patients will have 45 minutes of progressive therapeutic exercise training (PTE) with the telerehabilitation method.
  Interventions: Behavioral: Progressive therapeutic exercise training
- Control Group (No Intervention): Group 3: Participants will be taken for the waiting list after evaluation with the telerehabilitation method.

INTERVENTIONS:
Behavioral: Pain Neuroscience education + Progressive therapeutic exercise training — The education group will have a comprehensive patient education which includes; description, transmission, representation of pain, central sensitization, neuroplasticity, its relation to body systems, psychosocial and emotional factors affecting pain, pain behavior, and lifestyle changes to cope with pain, etc. Plus, the group will have supervised progressive therapeutic exercises via the telerehabilitation method.
  Arms: Education+Exercise Group
Behavioral: Progressive therapeutic exercise training — The exercise group will have supervised progressive therapeutic exercises via the telerehabilitation method.
  Arms: Exercise group

SUMMARY:
The study investigates the effects of pain and exercise training via telerehabilitation method on pain, pain beliefs, trunk mobility, functionality, and quality of life in individuals with low back pain caused by facet joint arthrosis. Forty - five individuals are planning to include in the study. Participants will be randomly assigned to one of the three groups: Group 1: Pain education + exercise training group, Group 2: Exercise training group, and Group 3: Control group. The same physiotherapist will make evaluations via an online conference system. Group 1 will have pain neuroscience education and progressive therapeutic exercise training in a session for six weeks, twice a week, and Group 2 will have progressive therapeutic exercise training in a session for six weeks, twice a week, for six weeks, in total twelve sessions. Group 3 participants will be taken to the waiting list. Clinical and demographic data of the 45 participants in the study will be taken pre and post interventions. The primary outcomes are; the Numeric Pain Rating Scale (NPRS) and the Oswestry Disability Index (ODI). Secondary outcomes are the Active Straight Leg Raise Test (A- SLR), The Pain Belief Questionnaire (PBQ), and the Short Form Quality of Life Form (SF-12). Statistical analysis will be run through the SPSS 20.0 package program.

DETAILED DESCRIPTION:
'Pain Neuroscience Education (PNE) is one of the cognitive approaches among conservative treatments, and has been one of the most inquisitive approaches. The content of the education includes the physiology of pain, types of pain, the areas in which it is represented in the brain, its effect on body image, and psychosocial dimensions. Education aims to break the patient's misinformation and perception about pain and teach how to manage pain. It aims to inform patients about the neurophysiological and neurobiological processes related to the pain experience and help change their misinformation about pain conditions. Improved pain knowledge changes attitudes and beliefs about pain, reduces destructive thoughts, and fear of pain, and improves physical performance. It is known to reduce pain and disability according to short-term results in patients with chronic pain with central sensitization. According to systematic reviews, PNE is moderately effective in patients with chronic musculoskeletal pain. In addition, it is stated that the use of educational approaches based on the neurophysiology of pain offers clinical benefits not only in physical terms but also in psychosocial terms. Since maladaptive psychosocial factors (for example, negative emotions, poor self-efficacy, and maladaptive beliefs) are associated with pain behaviors, it is thought that increasing pain knowledge will have an impact on pain perception. In a study conducted on patients with musculoskeletal pain who experience different types of pain, an inverse relationship between pain intensity and knowledge level was shown.

Due to the COVID-19 pandemic, the interest in the telerehabilitation method has increased, and it has become reachable easier with more evidence value on this subject. However, physiotherapists are healthcare professionals who work face-to-face with patients; depending on the pandemic curfews, the World Health Organization (WHO) has recommended not to continue face-to-face practices, except in emergencies, to protect patients' and physiotherapists' health. While digital options such as sensors, wearable technologies, virtual reality, and artificial intelligence are considered a solution, Tele-Rehabilitation (TR) can be the most practical, reachable, and cheaper solution to existing problems.

Systematic research and meta-analyses examining the effect of the telerehabilitation method and comparing it with traditional rehabilitation have revealed similar gains in outcome measures such as pain intensity and quality of life. It has been reported that simultaneous TR has comparable and effective results with face-to-face rehabilitation on pain and function in musculoskeletal problems. The telerehabilitation method is effective and cost-effective, especially in low back pain. Revealing the effects with more specific patient groups is the common recommendation of the studies.

In line with this information, the study's primary purpose is to determine the effects of PNE and progressive therapeutic exercise training given by the physiotherapist with the telerehabilitation method on pain, disability, pain beliefs, and quality of life. The secondary aim is to compare the effectiveness of progressive therapeutic exercise training alone or with PNE.

ELIGIBILITY:
Inclusion Criteria:

* volunteering,
* being the ages of 40 to 64
* having a diagnosis of Grade 1 or 2 facet joint arthrosis according to Pathria classification
* having pain for at least 12 weeks, primarily due to facet joint arthrosis
* having a pain score between 3 and 8 according to the Numerical Pain Scale (NRS)
* not having received education about pain before,
* having computer and internet access

Exclusion Criteria:

* having a BMI of 30 and above
* to have had conservative treatment or surgery in the lumbar region in the last 6 months,
* having severe deformity in the lower extremity
* having red or orange (pregnancy, disc pathology, infection, fracture, cancer, stenosis, severe osteoporosis, schmorl nodule, cauda equina syndrome, etc.) signs defined for low back pain
* having a regular exercise habit,
* having a seronegative rheumatological disease,
* having general pain syndrome.

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
The Numerical Rating Scale | Pre - intervention
  It is a frequently used scale with proven validity and reliability (Clark 2003, Boonstra 2008), consists of a horizontal line 100 mm long. There are two marks at the beginning and end of the line. The mark at the beginning of the line indicates 0 mm - no pain; the mark at the end of the line - 100 mm - unbearable pain. Subjects will be asked to place a mark on this horizontal line for the maximum pain they feel during rest and activity, and the results will be recorded in cm.
The Numerical Rating Scale | 6 weeks later (Post intervention)
  It is a frequently used scale with proven validity and reliability (Clark 2003, Boonstra 2008), consists of a horizontal line 100 mm long. There are two marks at the beginning and end of the line. The mark at the beginning of the line indicates 0 mm - no pain; the mark at the end of the line - 100 mm - unbearable pain. Subjects will be asked to place a mark on this horizontal line for the maximum pain they feel during rest and activity, and the results will be recorded in cm.
The Oswestry Disability Index | Pre - intervention
  The Oswestry Disability Index(ODI) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools. Scores between 0-5 are given for each question on the scale consisting of 10 questions. Questions are on travel, social life, sex life, sleeping, standing, sitting, walking, lifting things and personal precautions. Maximum score is 50, minimum score is 0.
The Oswestry Disability Index | 6 weeks later (Post intervention)
  The Oswestry Disability Index(ODI) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools. Scores between 0-5 are given for each question on the scale consisting of 10 questions. Questions are on travel, social life, sex life, sleeping, standing, sitting, walking, lifting things and personal precautions. Maximum score is 50, minimum score is 0.

SECONDARY OUTCOMES:
Active Straight Leg Raise Test | Pre - intervention
  The ASLR test was performed with the patient in a supine position with straight legs and feet 20 cm apart. The first instruction to the patient was "Try to raise your legs, one after the other, above the couch 20 cm without bending the knee." The patient was asked to score impairment on a 6-point scale with the following choice options: 0 (not difficult at all), 1 (minimally difficult), 2 (somewhat difficult), 3 (fairly difficult), 4 (very difficult), 5 (unable to perform). The scores of both sides were added, with the summed score ranging from 0 to 10.
Active Straight Leg Raise Test | 6 weeks later (Post intervention)
  The ASLR test was performed with the patient in a supine position with straight legs and feet 20 cm apart. The first instruction to the patient was "Try to raise your legs, one after the other, above the couch 20 cm without bending the knee." The patient was asked to score impairment on a 6-point scale with the following choice options: 0 (not difficult at all), 1 (minimally difficult), 2 (somewhat difficult), 3 (fairly difficult), 4 (very difficult), 5 (unable to perform). The scores of both sides were added, with the summed score ranging from 0 to 10.
The Short Form 12 | Pre - intervention
  It is a 12-item scale that evaluates the health-related quality of life, consisting of 8 sub-parameters, including physical function, physical role difficulty, pain, general health, vitality, social function, emotional role difficulty, and mental status (Ware 1994, Demiral 2006). It is scored between 0 and 100; the higher the score, the better quality of life.
The Short Form 12 | 6 weeks later (Post intervention)
  It is a 12-item scale that evaluates the health-related quality of life, consisting of 8 sub-parameters, including physical function, physical role difficulty, pain, general health, vitality, social function, emotional role difficulty, and mental status (Ware 1994, Demiral 2006). It is scored between 0 and 100; the higher the score, the better quality of life.
The Pain Beliefs Questionnaire | Pre - intervention
  Edwards et al. in 1992 developed to evaluate beliefs about the cause and treatment of pain (Edwards et al. 1992), validity in Turkish patients, and reliability study of the scale was conducted by Berk in 2006 (Berk, 2006). There are 12 items on this scale covering pain beliefs. Accordingly, it consisted of two test areas: Organic Beliefs consisting of 8 items and Psychological Beliefs consisting of 4 items. There is no cut-off point in the score. As the score increased, the internal consistency scores were measured with the Cronbach Alpha coefficient and reported as 0.71 for the Organic Beliefs subtest and 0.73 for the Psychological Beliefs subtest. The patient is asked to mark the most appropriate one for each item from 6 Likert-type options between 1: never and 6: always. The score for each subtest is calculated by adding the scores obtained from the items and dividing the number of items.
The Pain Beliefs Questionnaire | 6 weeks later (Post intervention)
  Edwards et al. in 1992 developed to evaluate beliefs about the cause and treatment of pain (Edwards et al. 1992), validity in Turkish patients, and reliability study of the scale was conducted by Berk in 2006 (Berk, 2006). There are 12 items on this scale covering pain beliefs. Accordingly, it consisted of two test areas: Organic Beliefs consisting of 8 items and Psychological Beliefs consisting of 4 items. There is no cut-off point in the score. As the score increased, the internal consistency scores were measured with the Cronbach Alpha coefficient and reported as 0.71 for the Organic Beliefs subtest and 0.73 for the Psychological Beliefs subtest. The patient is asked to mark the most appropriate one for each item from 6 Likert-type options between 1: never and 6: always. The score for each subtest is calculated by adding the scores obtained from the items and dividing the number of items.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University - Cerrahpaşa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Clarke CL, Ryan CG, Martin DJ. Pain neurophysiology education for the management of individuals with chronic low back pain: systematic review and meta-analysis. Man Ther. 2011 Dec;16(6):544-9. doi: 10.1016/j.math.2011.05.003. Epub 2011 Jun 25. PMID 21705261
- [Background] Cottrell MA, Galea OA, O'Leary SP, Hill AJ, Russell TG. Real-time telerehabilitation for the treatment of musculoskeletal conditions is effective and comparable to standard practice: a systematic review and meta-analysis. Clin Rehabil. 2017 May;31(5):625-638. doi: 10.1177/0269215516645148. Epub 2016 May 2. PMID 27141087
- [Background] Fatoye F, Gebrye T, Fatoye C, Mbada CE, Olaoye MI, Odole AC, Dada O. The Clinical and Cost-Effectiveness of Telerehabilitation for People With Nonspecific Chronic Low Back Pain: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Jun 24;8(6):e15375. doi: 10.2196/15375. PMID 32357128
- [Background] Louw A, Diener I, Butler DS, Puentedura EJ. The effect of neuroscience education on pain, disability, anxiety, and stress in chronic musculoskeletal pain. Arch Phys Med Rehabil. 2011 Dec;92(12):2041-56. doi: 10.1016/j.apmr.2011.07.198. PMID 22133255
- [Background] Louw A, Zimney K, Puentedura EJ, Diener I. The efficacy of pain neuroscience education on musculoskeletal pain: A systematic review of the literature. Physiother Theory Pract. 2016 Jul;32(5):332-55. doi: 10.1080/09593985.2016.1194646. Epub 2016 Jun 28. PMID 27351541
- [Background] Moseley L. Combined physiotherapy and education is efficacious for chronic low back pain. Aust J Physiother. 2002;48(4):297-302. doi: 10.1016/s0004-9514(14)60169-0. PMID 12443524
- [Background] Palacin-Marin F, Esteban-Moreno B, Olea N, Herrera-Viedma E, Arroyo-Morales M. Agreement between telerehabilitation and face-to-face clinical outcome assessments for low back pain in primary care. Spine (Phila Pa 1976). 2013 May 15;38(11):947-52. doi: 10.1097/BRS.0b013e318281a36c. PMID 23238489
- [Background] Bodes Pardo G, Lluch Girbes E, Roussel NA, Gallego Izquierdo T, Jimenez Penick V, Pecos Martin D. Pain Neurophysiology Education and Therapeutic Exercise for Patients With Chronic Low Back Pain: A Single-Blind Randomized Controlled Trial. Arch Phys Med Rehabil. 2018 Feb;99(2):338-347. doi: 10.1016/j.apmr.2017.10.016. Epub 2017 Nov 11. PMID 29138049
- [Background] Saracoglu I, Arik MI, Afsar E, Gokpinar HH. The effectiveness of pain neuroscience education combined with manual therapy and home exercise for chronic low back pain: A single-blind randomized controlled trial. Physiother Theory Pract. 2022 Jul;38(7):868-878. doi: 10.1080/09593985.2020.1809046. Epub 2020 Aug 19. PMID 32812478
- [Background] Truter P, Russell T, Fary R. The validity of physical therapy assessment of low back pain via telerehabilitation in a clinical setting. Telemed J E Health. 2014 Feb;20(2):161-7. doi: 10.1089/tmj.2013.0088. Epub 2013 Nov 27. PMID 24283249
- [Background] Turolla A, Rossettini G, Viceconti A, Palese A, Geri T. Musculoskeletal Physical Therapy During the COVID-19 Pandemic: Is Telerehabilitation the Answer? Phys Ther. 2020 Aug 12;100(8):1260-1264. doi: 10.1093/ptj/pzaa093. No abstract available. PMID 32386218
- [Background] Wood L, Hendrick PA. A systematic review and meta-analysis of pain neuroscience education for chronic low back pain: Short-and long-term outcomes of pain and disability. Eur J Pain. 2019 Feb;23(2):234-249. doi: 10.1002/ejp.1314. Epub 2018 Oct 14. PMID 30178503
- [Derived] Tahran O, Ersoz Huseyinsinoglu B, Yolcu G, Karadag Saygi E, Yeldan I. Comparing face-to-face and internet-based basic body awareness therapy for fibromyalgia: a randomized controlled trial. Disabil Rehabil. 2025 Sep;47(19):4987-4998. doi: 10.1080/09638288.2025.2465597. Epub 2025 Feb 19. PMID 39970076
- See also: Application — https://play.google.com/store/apps/details?id=com.drinkplusplus.angle&hl=en_US&gl=US
- See also: WCPT — https://www.wcpt.org/news/report-sets-out-future-of-digital-physical-therapy-practice